CLINICAL TRIAL: NCT05247580
Title: Impact Assessment of an Interdisciplinary and Multimodal Hospital Program of Pediatric Medical Emergencies' in Situ Simulation
Brief Title: Impact of Pediatric Medical Emergencies' in Situ Simulations
Acronym: Impact-SUrVIS
Status: Withdrawn | Type: Observational
Why Stopped: The manager could not start the search.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211546
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pedagogical and Psycho-social Impact of in Situ Simulation
Keywords: Hospital healthcare simulation program; Pediatric medical emergencies; Cross-cutting skills; Communication skills; Human factors; Self-confidence; Teamwork; Team leading; Work-related stress
MeSH Terms: conditions — Occupational Stress | interventions — Maslach Burnout Inventory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospital staff caregivers: Necker - Enfants Malades hospital' nurses, nurses' aides, residents and, doctors of medicine.
  Interventions: Other: Hicks self-confidence scale, Karasek survey, Maslach Burnout Inventory

INTERVENTIONS:
Other: Hicks self-confidence scale, Karasek survey, Maslach Burnout Inventory — Questionnaires (Hicks self-confidence scale, Karasek questionnaire, Maslach Burnout Inventory) sent to hospital staff caregivers before and after (at 3 and 6 months) their SUrVIS training.

SUMMARY:
Simulation in healthcare is becoming more and more essential in the training of paramedical and medical caregivers. It is a powerful educational tool that can enrich knowledge and skills, whether technical (setting up a venous catheter, intubation, etc...) or transversal (teamwork, communication, stress management in crises, etc.).

The hospital environment requires nurses, nurses' aides, residents, and doctors to provide human care in increasingly technical work environments while exercising increasing responsibilities. These caregivers are therefore exposed to many stressors. Several studies highlight the benefits of simulation on the ability of professionals to deal with rare and/or complex crises which they have previously faced during simulation sessions.

Beginning January 2022, the Necker - Enfants Malades hospital will start a hospital' scale training program for pediatric medical emergencies using in situ simulation of the Necker - Enfants Malades hospital.

The SUrVIS (Simulation d'Urgences Vitales In Situ) project is based on interprofessional training courses divided into four parts theoretical training (recognition of the critically ill child / cardiorespiratory arrest, how to call for assistance), procedural simulation (ventilation / chest compression / set up an intraosseous access / call for help...), three in situ simulation scenarios of pediatric medical emergencies (with live audiovisual retransmission for observers) each ending with a debriefing and a conclusion of the day with handing over of best practice documents. The study investigation team plan to train 400 caregivers each year (including 300 nurses and nurses' aides).

The Impact-SUrVIS (Impact de la Simulation d'Urgences Vitales In Situ) study is built around the SUrVIS sessions. Through questionnaire, the study investigation team will assess the impact of this hospital program on self-confidence, the feeling of professional efficiency, interprofessional communication, and work-related stress.

DETAILED DESCRIPTION:
The SUrVIS project is structured around a 12-persons one-day interdisciplinary in situ simulation training sessions including:

* Training in...

  * Recognition of the critically ill child and pediatric cardiopulmonary arrest
  * The call for help according to the SAED method (Haute Autorité de Santé)
  * Interprofessional communication and human factors in healthcare
* Procedural simulation workshops: intraosseous line placement, bag-mask ventilation, emergency drugs preparation, call for help simulations...
* Three 4-persons in situ simulation scenarios of pediatric medical emergencies (e.g., cardiorespiratory arrest, acute respiratory failure, arrhythmias, cardiogenic shock, status epilepticus, pediatric polytrauma, medical emergency during a surgery...), with live audiovisual retransmission for the 8 learners not participating in the scenario. Each scenario will be followed by a 45' debriefing with all learners in a dedicated room. Scenarios will also be built around adverse events in healthcare previously analyzed in a Morbidity Mortality Review (MMR). The constitution of a small group (12 persons) allows all learners to participate at least once in the scenarios (unless one or more learners wish otherwise).
* A conclusion of the day and a hand-over of cognitive aids created by the management team.

Twelve trainees, 1/4 of whom are physicians or residents and 3/4 of whom are nurses or nursing assistants, will participate in each SUrVIS session.

All the in situ simulation scenarios will take place in the Necker - Enfants Malades Hospital departments (general pediatrics, pediatric nephrology, etc.). The main objective is to increase the psychological fidelity of these training sessions. Indeed, the learners will practice in familiar environments with the material of their daily practice. After the training day, the training team will remain at the disposal of the learners for an individual debriefing if they wish.

The Impact-SUrVIS study is built around the SUrVIS sessions. Through questionnaires, the study investigation team will assess the impact of our program. The study investigation team will send the participating nurses, nurses' aides, residents and doctors a pre-test questionnaire, based on standardized scales. Then the study investigation team will carry out a post-test re-evaluation at 3 and 6 months.

The main objective of the Impact-SUrVIS study is to evaluate the effects of the SUrVIS program on pediatric medical emergencies management self-confidence using the Hicks Self-Confidence Scale.

The secondary objectives of the Impact-SUrVIS study are to:

* Study the beneficial effects of the SUrVIS program on psychological demand, decision latitude, and social support using the Karasek survey.
* Study the impact of the SUrVIS program on the quality of life at work (work-related stress, burnout) using the Maslach Burnout Inventory.

ELIGIBILITY:
Inclusion Criteria:

1. Any caregivers staff at Necker - Enfants Malades Hospital agreeing to participate in the Impact-SUrVIS study and thoroughly complete the Impact-SUrVIS study questionnaires.
2. Non-medical staff at Necker - Enfants Malades Hospital:

   * Attending nurses
   * Attending nurses' aides
   * Student nurse
   * Student nurses' aides
3. Medical staff at Necker - Enfants Malades Hospital:

   * Doctor of Medicine (M.D.)
   * Pediatrics, Emergency Medicine and Anesthesia/Intensive care Residents.

Exclusion Criteria:

Medical student

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers staff at Necker - Enfants Malades Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Feeling of professional efficiency | 6 months
  Evaluate the effects of the SUrVIS program on pediatric medical emergencies management self-confidence using the Hicks Self-Confidence Scale.
  The Hicks self-confidence scale is a Likert-type self-confidence scale (Hicks, 2006) consisting of 12 items was created to measure this variable. The response option of each item ranges from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicating greater self-confidence.

SECONDARY OUTCOMES:
Psychological demand, decision latitude, and social support | 6 months
  Study the beneficial effects of the SUrVIS program on psychological demand, decision latitude, and social support using the Karasek questionnaire.
  This questionnaire evaluates three dimensions of the psychosocial work environment: psychological demand, decision latitude, and social support. It includes 26 questions: nine for psychological demand, nine for decision latitude, and eight for social support. The proposed answers are: "Strongly disagree," "Disagree," "Agree," and "Strongly agree," which makes it possible to rate them from 1 to 4 and to calculate a score for each of the three dimensions. Then the median value of each score will be calculated, i.e., the value dividing the entire surveyed population into two equal parts: half are above this score, and the other half are below it. Job strain is defined as a situation where psychological demand is above the median and decision latitude is below the median, which constitutes a health-risk situation.
Work-related stress and burnout | 6 months
  Study the impact of the SUrVIS program on the quality of life at work (work-related stress, burnout) using the Maslach Burnout Inventory (MBI)
  The MBI is a 22-item frequency scale representing the three dimensions of burnout:
  * Emotional exhaustion (EE)
  * Depersonalization (DP) OR Dehumanization
  * Loss of personal accomplishment (PA) For each dimension: " low", " moderate ", " high " score. A high score of (EE) or (DP) OR a low score of (PA) is sufficient to speak of burnout.
  Depending on the number of dimensions affected, there are stages of severity. The degree of burnout is said to be:
  * Low: only one dimension is affected.
  * Medium: two out of three dimensions are affected.
  * Severe: all three dimensions are pathological.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu BENDAVID, M.D., Principal Investigator — Assistance Publique - Hôpitaux de Paris; Sylvain RENOLLEAU, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No